CLINICAL TRIAL: NCT01623700
Title: A Retrospective Epidemiological Study to Investigate Outcome and Mortality With Longterm Antithrombotic Therapy in Acute Coronary Syndrome Patients
Brief Title: Outcome of Longterm Antithrombotic Therapy in Acute Coronary Syndrome Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uppsala University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: U-11-001
Record Dates: First submitted 2012-05-29; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2011-05

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction
Keywords: clopidogrel; aspirin; percutaneous coronary intervention; coronary stenting; antiplatelet
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- dual antiplatelet treatment 12 months after ACS event
- dual antiplatelet treatment 6 months after ACS event
- dual antiplatelet treatment 3 months after ACS event

SUMMARY:
This observational study will based on the Register of Information and Knowledge About Swedish Heart Intensive Care Admissions (RIKS-HIA) and the Swedish Coronary Angiography and Angioplasty Registry (SCAAR) which since 2009 are merged into The Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART).

The aim of this study is to investigate the impact of different antithrombotic treatment options (treatment duration, type of treatment and combination of treatments) in Acute Coronary Syndrome (ACS) patients on outcomes such as recurrent ischemic events and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an event of ACS under the study period
* Patient found in the National Registry of Drug Prescriptions and treated or not treated with antithrombotic drug/s (acetylsalicylic acid and/or either clopidogrel/ticlopidine/prasugrel and/or warfarin)

Exclusion Criteria:

* Patients will not be excluded from the database if they fulfill inclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients previously enrolled into the SWEDEHEART (RIKS-HIA/SCAAR/SEPHIA) registry from 1 Jan 2006 to 1 July 2010 with an event of ACS and observed during the index hospitalization following enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 78000 (Actual)
Dates: Start 2006-01

PRIMARY OUTCOMES:
number of patients with adverse events in patient groups with different antithrombotic treatment strategies | up to 5 years and 6 months
  adverse events such as: mortality, re-infarction, revascularization, ischemic- and non-ischemic stroke and bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Stefan James, MD, PhD, Principal Investigator — Uppsala Clinical Research Center and Department of Medical Sciences, Cardiology
Locations (1):
- Uppsala Clinical Research Center and Department of Medical Sciences, Uppsala University, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Varenhorst C, Jensevik K, Jernberg T, Sundstrom A, Hasvold P, Held C, Lagerqvist B, James S. Duration of dual antiplatelet treatment with clopidogrel and aspirin in patients with acute coronary syndrome. Eur Heart J. 2014 Apr;35(15):969-78. doi: 10.1093/eurheartj/eht438. Epub 2013 Oct 11. PMID 24122961